CLINICAL TRIAL: NCT01466205
Title: Clinical Testing of a D1 Agonist for Cognitive Enhancement in Schizotypal Personality Disorder
Acronym: SPD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Larry J. Siever (Other)
Collaborators: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor-Investigator, Larry J. Siever, Executive Director, Mental Illness Research Education and Clinical Center (MIRECC); Chief, Psychiatry Program, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-0110
Record Dates: First submitted 2011-10-27; First posted 2011-11-07 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Cognitive Impairments; Schizotypal Personality Disorder
Keywords: schizotypal personality disorder; cognitive impairment; working memory
MeSH Terms: conditions — Cognitive Dysfunction; Schizotypal Personality Disorder | interventions — dihydrexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DAR 0-100A (Experimental): The examination of SPD subjects, who are more likely than schizophrenia patients to show significant cognitive improvement after the use of single doses of dopamine agonists, such as DAR-0100A provides an excellent opportunity to demonstrate the effectiveness of D1 agonists on cognition in the schizophrenia spectrum.
  Interventions: Drug: DAR-0100A
- Placebo (Placebo Comparator): Some subjects receive placebo, instead of the study drug, in a double-blind randomized fashion. This allows for performance comparison between SPD subjects on DAR-0100A and those on placebo. The hypothesis is that SPD subjects on DAR-100A will show improvement on primary measures greater than SPD subjects randomized to placebo between baseline and post-drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DAR-0100A — DAR-0100A will be administered intravenously in a dose of 15mg in 150mls of saline over 30 minutes at approximately 11:00AM on each of three consecutive days of administration. Additional saline will be co-administered to ensure hydration.
  Arms: DAR 0-100A
Drug: Placebo — 150mls of saline is administered over 30 minutes at approximately 11:00AM on each of three consecutive days of administration. Additional saline will be co-administered to ensure hydration.
  Arms: Placebo

SUMMARY:
Currently, no study to date has directly tested a selective D1R agonist in relation to the cognitive impairment of Schizophrenia without the confound of neuroleptics. The investigators propose to examine the efficacy of DAR-0100A, a highly selective, full D1R agonist supported by pre-clinical and preliminary pilot clinical data, in ameliorating the cognitive deficits in Schizotypal Personality Disordered subjects receiving no medications including antipsychotics.

The investigators hypothesize that 1) Baseline primary outcome measures will be impaired in Schizotypal personality disorder (SPD) subjects compared to controls, 2) SPD subjects on DAR-0100A will show improvement on primary measures greater than healthy controls and SPD patients randomized to placebo, and 3) SPD patients will show significant improvements on primary outcome variables on drug compared to placebo.

DETAILED DESCRIPTION:
Working memory deficits are central to the cognitive impairment of schizophrenia and other psychiatric disorders. The D1 receptor (D1R) is probably the best established mediator of working memory in neuroscience studies for over three decades and represents a highly promising therapeutic target for enhancing working memory in these disorders, yet this mechanism has never been tested in humans. Schizotypal personality disorder (SPD) patients who evidence moderate, focal impairments in working memory represent a unique population to test the effect of a D1 agonist on working memory impairment in humans. Cognitive impairment is the most salient predictor of functional outcome in schizophrenia (SCZ) and is essentially refractory to conventional treatments. Identifying pharmacologic agents that target the cognitive deficits of SCZ is thus the top priority in SCZ research, but so far, clinical trials of a number of drugs with preclinical promise have yielded disappointing results. Currently, no study to date has directly tested a selective D1R agonist in relation to the cognitive impairment of SCZ without the confound of neuroleptics. The investigators propose to examine the efficacy of DAR-0100A, a highly selective, full D1R agonist supported by pre-clinical and preliminary pilot clinical data, in ameliorating the cognitive deficits in SPD subjects receiving no medications including antipsychotics. SPD will be classified as a schizophrenic disorder in DSM-5 and ICD-10. The investigators have characterized the cognitive deficits of SPD and demonstrated that, as with chronic SCZ, a core component consists of impairments in working memory. Studies of SPD obviate confounds associated with SCZ, such as the effects of overt psychotic episodes, medication history, severe, persistent functional impairment and multiple treatments. Furthermore, the cognitive deficits of SPD are less global and more readily reversible than those of chronic SCZ, providing a unique opportunity to test the D1 mechanism of cognitive enhancement. DAR-0100A, which is the active enantiomer of dihydrexidine (DHX), is a full D1R agonist with a10-60 fold selectivity over the D2R. DHX administration improves cognition in single doses in young adult and aged monkeys and rodents. A single treatment with DAR-0100A in adult humans with SCZ was demonstrated to enhance prefrontal perfusion. Pilot data from our group and Columbia suggest DAR-0100A improves cognitive performance, particularly working memory, in the schizophrenia spectrum.

Primary Aims: 1. To perform a 5-year study in which three consecutive days of DAR-0100A at a dose of 15 mg or placebo are administered intravenously over 30 minutes to 60 patients with SPD (12/yr) in a between-groups, randomized, double-blind design. Cognitive testing will be performed at baseline (Day 1) and on the third day of drug/placebo administration (Day 4). Subjects will return at Day 15 to receive drug (if randomized initially to placebo) or placebo (if randomized to drug) in a double blind fashion in an identical protocol. This allows all patients to receive drug for Secondary Aim 1 while maintaining the blind. Baseline (Day 1) and repeat cognitive testing (Day 4) is also administered to 60 healthy controls per year (12/yr). The cognitive tests of working memory serving as primary outcome measures will include the modified AX-CPT (d'), the N-back (% correct at the 2-back condition), the DOT Task (distance error at 30 second delay - no delay), and the Paced Auditory Serial Addition Task (PASAT)( correct responses). The investigators will also include other tests of memory, executive function, and verbal learning for secondary outcome measures (see Methods) as well as comparison tests not hypothesized to change with drug: the Benton line orientation test (JLOT) and the Trail Making Test A. 2. To compare changes on the primary outcome measures from baseline to Day 4 testing between drug and placebo administration in SPD subjects. 3. To compare primary outcome variables at baseline and change from baseline to Day 4 testing between patients groups and healthy controls. 4. To obtain plasma DHX concentrations on Day 4 to evaluate plasma concentrations in relation to cognitive changes as a potential covariate.

Secondary Aims: 1. To evaluate the change between baseline and Day 4 cognitive testing in all SPD patients receiving drug in the first or second phase. 2. To evaluate secondary outcome and comparison variables between SPD patients on placebo and drug.

Primary Hypotheses: 1. Baseline primary outcome measures will be impaired in SPD subjects compared to controls. 2. SPD subjects on DAR-0100A will show improvement on primary measures greater than healthy controls and SPD patients randomized to placebo between baseline and Day 4. 3. SPD patients will show significant improvements on primary outcome variables on drug compared to placebo but not on comparis¬on perceptual (JLOT) and processing speed/attentional tasks (Trails A).

It is critical to establish efficacy for cognitive enhancement with a selective D1 agonist in a schizophrenic disorder with cognitive impairment and without concomitant neuroleptic treatment to provide momentum for these efforts. The more readily reversible cognitive impairment of SPD provides a unique opportunity for this critical study of the D1 hypothesis to pave the way for development for more severe schizophrenic disorders with their inevitable complicating artifacts.

ELIGIBILITY:
Inclusion Criteria:

* Currently meeting DSM-IV-TR criteria for Schizotypal Personality Disorder
* Males and Females 18 ≤ age ≤ 60
* Medically and neurologically healthy
* Willing and having capacity to provide informed consent

Exclusion Criteria:

* Currently bipolar I disorder, schizophrenia or current psychosis
* Clinically significant cardiovascular or neurological conditions, uncontrolled hypertension, clinically significant EKG abnormalities, or serious general medical illness
* Clinical evidence of dehydration or significant hypotension
* Currently meeting DSM-IV-TR criteria for Major Depressive Disorder
* Current substance abuse or past dependence within the last six months (other than nicotine)
* Currently taking psychotropic medications
* Currently pregnant or lactating
* Non-English speaking

Socio-economically disadvantaged people will be included in our research study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of a D1 Agonist for Cognitive Enhancement of Working Memory in Schizotypal Personality Disorder | Baseline performance
  The cognitive tests of working memory serving as primary outcome measures will include the modified AX-CPT (d'), the N-Back (% correct at the 2-back condition), the DOT Task (distance error at 30 second delay--no delay), and the Paced Auditory Serial Addition Task (PASAT)(correct responses).
Efficacy of a D1 Agonist for Cognitive Enhancement of Working Memory in Schizotypal Personality Disorder | day one of drug administration
  The cognitive tests of working memory serving as primary outcome measures will include the modified AX-CPT (d'), the N-Back (% correct at the 2-back condition), the DOT Task (distance error at 30 second delay--no delay), and the Paced Auditory Serial Addition Task (PASAT)(correct responses).
Efficacy of a D1 Agonist for Cognitive Enhancement of Working Memory in Schizotypal Personality Disorder | after three days of drug administration
  The cognitive tests of working memory serving as primary outcome measures will include the modified AX-CPT (d'), the N-Back (% correct at the 2-back condition), the DOT Task (distance error at 30 second delay--no delay), and the Paced Auditory Serial Addition Task (PASAT)(correct responses).
Efficacy of a D1 Agonist for Cognitive Enhancement of Working Memory in Schizotypal Personality Disorder | one month after drug administration
  The cognitive tests of working memory serving as primary outcome measures will include the modified AX-CPT (d'), the N-Back (% correct at the 2-back condition), the DOT Task (distance error at 30 second delay--no delay), and the Paced Auditory Serial Addition Task (PASAT)(correct responses).

CONTACTS AND LOCATIONS:
Overall Officials: Larry J Siever, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Larry Siever, MD, Principal Investigator — James J Peters Bronx VA Hospital
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States